CLINICAL TRIAL: NCT01801488
Title: Genome-wide Analysis of Single Nucleotide Polymorphisms of Brain Arteriovenous Malformations and Cerebral Aneurysm
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#238810
Record Dates: First submitted 2012-12-12; First posted 2013-02-28 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2013-02

CONDITIONS: Arteriovenous Malformations; Intracranial Aneurysm; Subarachnoid Hemorrhage
MeSH Terms: conditions — Arteriovenous Malformations; Intracranial Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples of intracranial arterial-venous malformations (AVM) or aneurysm and blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AVM Patients: Patients receiving surgical intervention for an intracranial arterial-venous malformation.
- Ruptured Aneurysm: Patients receiving surgical intervention for a ruptured intracranial aneurysm.
- Unruptured Aneurysm: Patients receiving surgical intervention for an unruptured intracranial aneurysm.

SUMMARY:
Test single nucleotide polymorphisms (SNP's) in ruptured and unruptured aneurysm tissue to identify a genetic difference between the two types of aneurysms; and to test SNP's in arteriovenous malformation tissue to identify a genetic link.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients between the ages of 18 and 89 that are having open surgical resection of an AVM or clipping of an aneurysm will be included

Exclusion Criteria:

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to University Hospital.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Risk gene expression | Within one week of sample collection.
  The samples will be frozen after collection and then analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Deshaies, MD, Principal Investigator — SUNY Upstate Medical University Neurosurgery
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States